CLINICAL TRIAL: NCT06627569
Title: Exercise Effects on the Neurobiology Underlying Stress-Related Eating Behaviors in Veterans
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ENDA-009-24S; I01CX002752 (NIH)
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Overweight/Obesity; Stress
Keywords: Overweight; Obesity; Stress; Eating
MeSH Terms: conditions — Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be asked to complete 2 study days before and again after a 12-week intervention period, during which they will either continue with usual activities or be asked to complete exercise sessions four times per week. They will be randomly assigned to one of these conditions (exercise or not) and will not be able to choose their group assignment.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcomes assessors will not know the group assignment of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise (Experimental): Participants will complete 4 aerobic exercise training sessions per week for 12 weeks. The exercise program will begin at 15 minutes per session and duration will be gradually increased by 5 minutes each week until participants reach 30 minutes per session (with 5 min warm-up and cool-down). Exercise will be performed at a "moderate" intensity, which will be about 60-70% of your predicted maximal level. Participants will meet with study personnel once per week.
  Interventions: Behavioral: Exercise
- Usual activity (No Intervention): Participants will keep doing what they usually do for the 12-week intervention period. They will be asked not to change their usual physical activity levels during this period. They will meet with study personnel once per week

INTERVENTIONS:
Behavioral: Exercise — 12 weeks of aerobic exercise, with 4 sessions per week.
  Arms: Exercise

SUMMARY:
The purpose of this study is to learn more about how common lifestyle interventions, such as exercise, affect how our brains respond to performing thinking tasks and to viewing pictures of foods and various other objects. The investigators are also interested in how changes in hormones that might be different in men and women could affect how lifestyle interventions change these brain responses.

DETAILED DESCRIPTION:
The purpose of this study is to learn more about how common lifestyle interventions, such as exercise, affect how our brains respond to performing thinking tasks and to viewing pictures of foods and various other objects. The investigators are also interested in how changes in hormones that might be different in men and women could affect how lifestyle interventions change these brain responses. This will help us to better understand how different lifestyle interventions affect the brain and how this might relate to various behaviors. Eligible participants will be asked to complete 2 study days before and again after a 12-week intervention period, during which they will either continue with usual activities or be asked to complete exercise sessions four times per week. They will be randomly assigned to one of these conditions (exercise or not) and will not be able to choose their group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Veterans 18-75 years old
* BMI of 25 or greater
* Physically inactive
* Able to attend study visits in person in Aurora, CO

Exclusion Criteria:

* Currently pregnant
* History of bariatric surgery
* Current eating disorder
* Current treatment with appetite-altering medications (e.g., GLP-1 agonists)
* Contraindication to MRI (weight > 500 lbs; claustrophobia; metal or electronic devices in the body)
* Cardiovascular disease, chronic kidney disease, pulmonary disease, or diabetes
* Unable to exercise due to cardiac, pulmonary, neurologic, or orthopedic reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2030-08-30 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
Percent change in blood oxygen level dependent (BOLD) response to visual food cues as measured by functional magnetic resonance imaging (fMRI) | Baseline, 12 weeks
  Percent change in blood oxygen level dependent (BOLD) response from baseline to after the 12-week intervention period while viewing visual food cues. The primary contrast of interest is the comparison of high-calorie food images to nonfood object images.
Change in serum cortisol response to counting task | Baseline, 12 weeks
  Change from baseline to after the 12-week intervention period in serum cortisol levels (mcg/dL) throughout a counting task involving mental math (measured as area under the curve).

SECONDARY OUTCOMES:
Change in heart rate response to counting task | Baseline, 12 weeks
  Change from baseline to after the 12-week intervention period in heart rate (measured by photoplethysmograph; aggregated in 1 min intervals) throughout a counting task involving mental math (measured as area under the curve).

OTHER OUTCOMES:
Change in percent body fat | Baseline, 12 weeks
  Change in percent body fat, as measured by dual-energy x-ray absorptiometry, from baseline to after the 12-week intervention period.
Percent change in body weight | Baseline, 12 weeks
  Percent change in body weight (kg) from baseline to after the 12-week intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina T. Legget, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
As some journals now require authors to provide access to data, de-identified, anonymized data sets will be created after study results are published, and made available upon request for general research purposes, based on availability of resources. No proprietary data will be made publicly available. Sufficient data and descriptors will be made available to confirm conclusions in resulting publications and duplicate statistical analyses.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available after publication of study results and be available at least 3 years beyond the completion of the study.
Access Criteria: Data will be made available upon request for general research purposes, based on availability of resources.